CLINICAL TRIAL: NCT03977818
Title: Patterns of Care and Outcomes of Patients With METAstatic Soft Tissue SARComa in a Real-life Setting: the METASARC Observational Study
Brief Title: Patterns of Care and Outcomes in METAstatic Soft Tissue SARComa
Acronym: METASARC
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: French Sarcoma Group (Other)
Responsible Party: Sponsor
Other Study IDs: IB2017-METASARC
Record Dates: First submitted 2019-05-23; First posted 2019-06-06 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2020-12

CONDITIONS: Sarcoma; Metastases; Chemotherapy
Keywords: outcome; time to next treatment; overall survival; patterns of care
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with metastatic softtissue sarcomas diagnosed between 1990 and 2013

SUMMARY:
Well-designed observational studies of individuals with rare tumors are needed to improve patient care, clinical investigations, and the education of healthcare professionals.

The patterns of care, outcomes, and prognostic factors of a cohort of 2225 patients with metastatic soft tissue sarcomas who were diagnosed between 1990 and 2013 and documented in the prospectively maintained database of the French Sarcoma Group will be analyzed with a focus on : number/frequency of systemic treatments per patient, number/frequency of patients with locoregional treatment of the metastasis, number/frequency of patients with chemotherapy, number/frequency of patients with an off-label drug.

Outcome (time-to-next treatment [TNT] and overall survival [OS]) will be reported according to histological subtype, as well as the association between TNT and OS.

Prognostic factors of OS will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* advanced soft tissue sarcoma
* age > 18

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced soft tissue sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 2165 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, MD/PhD, Principal Investigator — Institut Bergonié, Comprehensive Cancer Center
Locations (3):
- France (3):
  - Institut Bergonié, Comprehensive Cancer Center, Bordeaux
  - Centre Léon Bérard, Comprehensive Cancer Center, Lyon
  - Institut Gustave Roussy, Comprehensive Cancer Center, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Savina M, Le Cesne A, Blay JY, Ray-Coquard I, Mir O, Toulmonde M, Cousin S, Terrier P, Ranchere-Vince D, Meeus P, Stoeckle E, Honore C, Sargos P, Sunyach MP, Le Pechoux C, Giraud A, Bellera C, Le Loarer F, Italiano A. Patterns of care and outcomes of patients with METAstatic soft tissue SARComa in a real-life setting: the METASARC observational study. BMC Med. 2017 Apr 10;15(1):78. doi: 10.1186/s12916-017-0831-7. PMID 28391775

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Metastatic Softtissue Sarcomas Diagnosed Between 1990 and 2013: Patients with metastatic softtissue sarcomas diagnosed between 1990 and 2013 and satisfying all eligibility criteria
Period: Overall Study
Arm/Group | Patients With Metastatic Softtissue Sarcomas Diagnosed Between 1990 and 2013
Started | 2165
Completed | 2165
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Metastatic Softtissue Sarcomas Diagnosed Between 1990 and 2013
Number analyzed (Participants) | 2165
Age, Customized [Count of Participants; unit: Participants]
  Age: < 75 years | 1886
  Age: >= 75 years | 279
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1110
  Male | 1055
Region of Enrollment [Number; unit: participants]
  France | 2165

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Time to Next Treatment (TNT) and Overall Survival (OS) Under First-line Treatment
Description: TNT: time from the systemic treatment onset to the next treatment or death due to any cause, whichever came first.
  OS: time from the systemic treatment onset to death
Time Frame: 2 years
Population: Patients with metastatic softtissue sarcomas diagnosed between 1990 and 2013 and satisfying all eligibility criteria
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Patients With Metastatic Softtissue Sarcomas Diagnosed Between 1990 and 2013
Number analyzed (Participants) | 2165
correlation coefficient | 0.76 [0.73 to 0.78]

ADVERSE EVENTS:
Groups:
- Patients With Metastatic Softtissue Sarcomas Diagnosed Between 1990 and 2013: Patients with metastatic softtissue sarcomas diagnosed between 1990 and 2013 satisfying all eligibility criteria
Arm/Group | Patients With Metastatic Softtissue Sarcomas Diagnosed Between 1990 and 2013
Serious Adverse Events (participants affected / at risk) | 0/2165
Other Adverse Events (participants affected / at risk) | 0/2165

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes